CLINICAL TRIAL: NCT03521583
Title: Von Willebrand Disease in the Netherlands - Prospective Study (WiN-Pro)
Brief Title: Von Willebrand Disease in the Netherlands
Acronym: WiN-Pro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Stichting Haemophilia (Dutch Haemophilia Foundation) (Unknown); CSL Behring (Industry); Shire (Industry)
Responsible Party: Principal Investigator, Frank W.G. Leebeek, MD, PhD, MD, PhD, Erasmus Medical Center
Other Study IDs: NL62238.078.18
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Von Willebrand Disease
Keywords: von Willebrand disease; von Willebrand factor; Nationwide study; Prospective study
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to prospectively investigate the current bleeding tendency of children and adults with VWD.

DETAILED DESCRIPTION:
Von Willebrand disease (VWD) is the most common inherited bleeding disorder, and is characterized by a defective platelet adhesion and aggregation. VWD is caused by a reduced (type 1), an abnormal function (type 2) or a complete absence (type 3) of von Willebrand factor (VWF).

In recent years, large retrospective cohort studies have provided valuable insights on the clinical presentation, bleeding phenotype, quality of life, diagnostics, genetics and treatment of patients with VWD. One of these large studies is the von Willebrand in the Netherlands (WiN) study, which is a nationwide cross sectional study of moderate and severe von Willebrand disease patients, that was initiated in 2007. Over 800 VWD patients were included in the WiN study, which was about 80% of all known VWD patients in the Netherlands. Although the WiN study and large retrospective studies in other countries provided important insights in understanding VWD, some significant challenges remain and large prospective studies are lacking to provide answers.

All large retrospective cohort studies have assessed the bleeding phenotype of patients with VWD using bleeding scores or retrospective questionnaires. Bleeding scores calculate the sum of all bleeding episodes during lifetime. Therefore, they provide useful information on the bleeding tendency during lifetime. However, bleeding scores do not provide information on the change of bleeding tendency. If a patient had a period in his or her lifetime in which he or she had many bleeding episodes, then the bleeding score is high. Though, the patient could have had those bleeds 30 years ago and did not have a bleeding episode since then. Therefore, bleeding scores do not provide information on the current bleeding phenotype of VWD patients. Furthermore, previous studies provided limited information on the frequency of mild bleedings, like gum bleeding or epistaxis, that occur in daily life but do not require therapy. Nevertheless, these bleeding episodes can cause a major impairment in quality of life. This is especially important in children, because school-going children with VWD have a lower quality of life and have a different bleeding tendency, characterized by more cutaneous bleeding (81%), oropharyngeal bleeding (64%) and epistaxis (56%).

Therefore, the primary aim of this study is to prospectively investigate the current bleeding tendency of children and adults with VWD.

ELIGIBILITY:
Inclusion Criteria:

* Historically lowest VWF:Ag and/or VWF:RCo and/or VWF:CB ≤ 0.30 IU/mL and/or FVIII:C ≤ 0.40 IU/mL
* Treatment at a Hemophilia treatment center in the Netherlands
* All types of VWD
* All ages

Exclusion Criteria:

- Other known bleeding disorders present.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Von Willebrand disease patients known in a Hemophilia Treatment Center in the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2019-07-28 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding rate | 2 years
  Number of bleedings in an individual divided by the follow-up duration

CONTACTS AND LOCATIONS:
Overall Officials: Frank WG Leebeek, MD, PhD, Principal Investigator — Erasmus Medical Center; Ferdows Atiq, MD, Study Director — Erasmus Medical Center; Marjon H Cnossen, MD, PhD, Study Chair — Erasmus Medical Center; Karin Fijnvandraat, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jeroen Eikenboom, MD, PhD, Study Chair — Leiden University Medical Center; Johanna G van der Bom, PhD, Study Chair — Leiden University Medical Center; Britta AP Laros-van Gorkom, MD, PhD, Study Chair — Radboud University Medical Center; Karina Meijer, MD, PhD, Study Chair — University Medical Center Groningen; Karin PM van Galen, MD, PhD, Study Chair — UMC Utrecht; Joke de Meris, Study Chair — Netherlands Hemophilia Society
Locations (9):
- Netherlands (9):
  - Academic Medical Center, Amsterdam
  - Maxima Medical Center, Eindhoven
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center +, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus University Medical Center, Rotterdam
  - Haga Hospital, The Hague
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leebeek FW, Eikenboom JC. Von Willebrand's Disease. N Engl J Med. 2016 Nov 24;375(21):2067-2080. doi: 10.1056/NEJMra1601561. No abstract available. PMID 27959741
- [Background] Sanders YV, Groeneveld D, Meijer K, Fijnvandraat K, Cnossen MH, van der Bom JG, Coppens M, de Meris J, Laros-van Gorkom BA, Mauser-Bunschoten EP, Leebeek FW, Eikenboom J; WiN study group. von Willebrand factor propeptide and the phenotypic classification of von Willebrand disease. Blood. 2015 May 7;125(19):3006-13. doi: 10.1182/blood-2014-09-603241. Epub 2015 Feb 11. PMID 25673639
- [Background] de Wee EM, Mauser-Bunschoten EP, Van Der Bom JG, Degenaar-Dujardin ME, Eikenboom HC, Fijnvandraat K, de Goede-Bolder A, Laros-van Gorkom BA, Meijer K, Raat H, Leebeek FW; Win Study Group. Health-related quality of life among adult patients with moderate and severe von Willebrand disease. J Thromb Haemost. 2010 Jul;8(7):1492-9. doi: 10.1111/j.1538-7836.2010.03864.x. Epub 2010 Mar 23. PMID 20345712
- [Background] de Wee EM, Sanders YV, Mauser-Bunschoten EP, van der Bom JG, Degenaar-Dujardin ME, Eikenboom J, de Goede-Bolder A, Laros-van Gorkom BA, Meijer K, Hamulyak K, Nijziel MR, Fijnvandraat K, Leebeek FW; WiN study group. Determinants of bleeding phenotype in adult patients with moderate or severe von Willebrand disease. Thromb Haemost. 2012 Oct;108(4):683-92. doi: 10.1160/TH12-04-0244. Epub 2012 Aug 23. PMID 22918553
- [Background] van Galen KPM, de Kleijn P, Foppen W, Eikenboom J, Meijer K, Schutgens REG, Fischer K, Cnossen MH, de Meris J, Fijnvandraat K, van der Bom JG, Laros-van Gorkom BAP, Leebeek FWG, Mauser-Bunschoten EP; Win study group. Long-term impact of joint bleeds in von Willebrand disease: a nested case-control study. Haematologica. 2017 Sep;102(9):1486-1493. doi: 10.3324/haematol.2017.168617. Epub 2017 Jun 1. PMID 28572165
- [Background] Sanders YV, Fijnvandraat K, Boender J, Mauser-Bunschoten EP, van der Bom JG, de Meris J, Smiers FJ, Granzen B, Brons P, Tamminga RY, Cnossen MH, Leebeek FW; WiN Study Group. Bleeding spectrum in children with moderate or severe von Willebrand disease: Relevance of pediatric-specific bleeding. Am J Hematol. 2015 Dec;90(12):1142-8. doi: 10.1002/ajh.24195. Epub 2015 Nov 17. PMID 26375306
- [Background] van Galen KPM, Meijer K, Vogely HC, Eikenboom J, Schutgens REG, Cnossen MH, Fijnvandraat K, van der Bom JG, Laros-van Gorkom BAP, Leebeek FWG, Mauser-Bunschoten EP; WiN study group. Joint surgery in von Willebrand disease: a multicentre cross-sectional study. Haemophilia. 2016 Mar;22(2):256-262. doi: 10.1111/hae.12834. Epub 2015 Nov 9. PMID 26551280
- [Background] Atiq F, Meijer K, Eikenboom J, Fijnvandraat K, Mauser-Bunschoten EP, van Galen KPM, Nijziel MR, Ypma PF, de Meris J, Laros-van Gorkom BAP, van der Bom JG, de Maat MP, Cnossen MH, Leebeek FWG; WiN study group. Comorbidities associated with higher von Willebrand factor (VWF) levels may explain the age-related increase of VWF in von Willebrand disease. Br J Haematol. 2018 Jul;182(1):93-105. doi: 10.1111/bjh.15277. Epub 2018 May 16. PMID 29767844